CLINICAL TRIAL: NCT01465308
Title: A Randomized Control Trial for the Effect of Honey on Radiotherapy Induced Xerostomia and Oral Mucositis in Patients With Head and Neck Cancers
Brief Title: The Effect of Honey on Xerostomia and Oral Mucositis
Acronym: AC-H
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cyprus University of Technology (Other)
Responsible Party: Principal Investigator, Dr. Andreas Charalambous, Lecturer-Researcher, Cyprus University of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AC-HANHS-86
Record Dates: First submitted 2011-10-31; First posted 2011-11-04 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer; radiotherapy induced xerostomia; radiotherapy induced oral mucositis; RCT; symptom management
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- receiving Honey (Experimental): The patients will receive honey mouthwash rinses
  Interventions: Dietary Supplement: Honey mouthwash
- Saline mouthwash (Active Comparator): The patients in this group will receive saline rinses
  Interventions: Other: Normal Saline

INTERVENTIONS:
Dietary Supplement: Honey mouthwash — The patients in the intervention group will receive honey mouthwash 15 minutes before the radiotherapy session, 15 minutes after and 6 hours after the radiotherapy session
  Arms: receiving Honey
Other: Normal Saline — Saline rinses 15 minutes before radiotherapy, 15 minutes after, and 6 hours after radiotherapy
  Arms: Saline mouthwash

SUMMARY:
The purpose of this study is to determine whether the use of pure honey will help in the treatment of radiation induced xerostomia and oral mucositis (symptom management)

DETAILED DESCRIPTION:
Radiation-induced mucositis is a normal acute side effect of radiotherapy treatment. Exposure of ionising radiation to oral, pharyngeal and laryngeal mucosa gives rise to radiation epithelitis towards the second and third weeks of conventional fractionated radiotherapy. Likewise, salivary flow may decrease by approximately 50% during the first week of radiotherapy and upwards of 80% by the seventh week of treatment. Acute radiation-induced xerostomia is associated with inflammatory reaction. The study will include an intervention and a control group, one receiving honey prior and after the radiotherapy and the other group not receiving honey at all.

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive radiotherapy (RT) to the oral cavity will be included in the study.
* Patients with a confirmed histologic diagnosis of head and neck cancer referred to non-palliative radiotherapy will enter into this trial.
* aged over 18
* receiving radiotherapy for at least four weeks

Exclusion Criteria:

* Allergic to honey
* confirmed and medically treated diabetes mellitus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-08; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Xerostomia grades | 1 week, 2 weeks, 3 weeks, 4 weeks
Change from baseline in oral mucositis grades | 1 week, 2 weeks, 3 weeks, 4 weeks

SECONDARY OUTCOMES:
Changes in the General satisfaction of comfort | 1 week, 2 week, 3 week, 4 week
Change in baseline weight in one month | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Charalambous, PhD, Principal Investigator — Cyprus University of Technology
Locations (1):
- Bank of Cyprus Oncology Centre, Nicosia, Nicosia, Cyprus

REFERENCES:
- [Derived] Charalambous M, Raftopoulos V, Paikousis L, Katodritis N, Lambrinou E, Vomvas D, Georgiou M, Charalambous A. The effect of the use of thyme honey in minimizing radiation - induced oral mucositis in head and neck cancer patients: A randomized controlled trial. Eur J Oncol Nurs. 2018 Jun;34:89-97. doi: 10.1016/j.ejon.2018.04.003. Epub 2018 Apr 30. PMID 29784145
- [Derived] Charalambous A, Lambrinou E, Katodritis N, Vomvas D, Raftopoulos V, Georgiou M, Paikousis L, Charalambous M. The effectiveness of thyme honey for the management of treatment-induced xerostomia in head and neck cancer patients: A feasibility randomized control trial. Eur J Oncol Nurs. 2017 Apr;27:1-8. doi: 10.1016/j.ejon.2017.01.001. Epub 2017 Jan 16. PMID 28279391